CLINICAL TRIAL: NCT06172920
Title: Comparison of the Analgesic Effects of Tramadol, Pethidine and Morphine Under Erector Spinae Plane (ESP) Block in the Treatment of Pain After Elective Thoracic Surgery
Brief Title: Comparison of Tramadol, Pethidine and Morphine in the Treatment of Pain After Thoracic Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Begüm Nemika Gökdemir, Begüm Nemika Gökdemir, Research Assistant of Anesthesiology Department, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KA23/137
Record Dates: First submitted 2023-10-10; First posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Thoracic Diseases; Analgesia
Keywords: thoracic surgery; patient controlled analgesia; postoperative care unit; intensive care
MeSH Terms: conditions — Thoracic Diseases; Agnosia | interventions — Tramadol

STUDY DESIGN:
Intervention Model Description: 3 groups of patients are received different type of analgesics
Who Masked: Participant, Care Provider
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tramadol (Active Comparator): Tramadol receiving group
  Interventions: Drug: Tramadol hydrochloride
- Aldolan (Active Comparator): Aldolan receiving group
  Interventions: Drug: Aldolan
- Morphine (Active Comparator): Morphine receiving group
  Interventions: Drug: Morphine hydrochloride

INTERVENTIONS:
Drug: Tramadol hydrochloride — Patients are receiving tramadol hydrochloride under thoracic surgery
  Arms: Tramadol
Drug: Aldolan — Patients are receiving meperidine under thoracic surgery
  Arms: Aldolan
Drug: Morphine hydrochloride — Patients are receiving Morphine hydrochloride under thoracic surgery
  Arms: Morphine

SUMMARY:
Comparison of analgesic effects of tramadol, aldolan and morphine under thoracic surgery

DETAILED DESCRIPTION:
Thoracotomy is one of the most painful surgical procedures known, and severe pain is encountered in 21-67% of patients after thoracotomy. The most important causes of this pain arise from the bone structures of the thoracic wall, damage to the costal joint junctions, stretching of the ligaments, rib fractures, and damage to the intercostal nerve and major muscles. Another factor that causes pain after thoracotomy is the chest tubes placed in the thorax to provide drainage (1).

As a result of this pain caused by loss of tissue and pulmonary reserve, effective coughing and decreased chest expansion can lead to serious complications such as atelectasis, ventilation/perfusion mismatch, hypoxemia, immobilization, thromboembolism and infection. These complications are associated with increased morbidity and mortality in thoracic surgery (2).

Ensuring pain management in patients undergoing thoracotomy is important in terms of reducing postoperative complications, ensuring early mobilization and increasing patient comfort. Since there is no single source that causes pain after thoracotomy, pain must be controlled at all levels. For this reason, a multimodal approach using pharmacological and non-pharmacological techniques is preferred in analgesia after thoracotomy. This approach reduces drug side effects along with the consumption of analgesics. Opioids and nonsteroidal anti-inflammatory drugs are used in pharmacological analgesia.

In our study, the investigators aim to compare the effects of tramadol, pethidine and morphine using intravenous patient-controlled analgesia in the treatment of postoperative pain in elective thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Having non-urgent thoracic surgery
* over 18 years old
* Being in group I-III according to the American Society of Anesthesiologists (ASA) classification
* Not have allergies to the drugs to be used (volunteers with diseases that prevent the use of drugs will not be included in the study
* regardless of gender

Exclusion Criteria:

. Have allergies to the drugs to be used

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-12-31 (Estimated); Primary Completion 2024-11-09 (Estimated); Study Completion 2024-12-09 (Estimated)

PRIMARY OUTCOMES:
The rate of drugs's analgesic effects | postoperative 24 hours
  To compare the analgesic effects of tramadol, pethidine and morphine in the treatment of postoperative pain in thoracic surgery, It will be assesed with numeric rating scale ( 0= no pain, 10= worst pain imaginable)
Comparing hemodynamic effects | Intraoperatively, then postoperative 24 hours
  To compare hemodynamic effects of tramadol, pethidine and morphine in the treatment of postoperative pain in thoracic surgery, It will be asssesed with measurements of intraoperative values of systolic, diastolic and mean arterial blood pressure
Comparing respiratory effects | postoperative 24 hours
  To compare respiratory effects of tramadol, pethidine and morphine in the treatment of postoperative pain in thoracic surgery. It will be asssesed with postoperative pulmonary complications such as failed extubation, bronchospasms or respiratory depressions.

SECONDARY OUTCOMES:
Adverse effects of analgesics | postoperative 24 hours
  It was aimed to compare the effects of drugs in terms of side effects, early mobilization.
surgeon satisfaction | Immediately after the surgery
  With a questionnaire, surgeon satisfaction will be assessed. (0 point= strongly disagree, 5 point= strongly agree)
patient satisfaction | Postoperative 30th minute
  With a questionnaire, patient satisfaction will be assessed. (0 point= strongly disagree, 5 point= strongly agree) When Aldrete score> 8, patient will be questioned for satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Baskent University Ankara Hospital, Ankara, Turkey (Türkiye)